CLINICAL TRIAL: NCT05717361
Title: The Effect of a Regimen of Opioid Sparing Anesthesia on Postoperative Recovery
Brief Title: Opioid Sparing Anesthesia in Cervical Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Evangelismos Hospital (Other)
Collaborators: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Athanasios Vaiopoulos, Anesthesia Resident, Evangelismos Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 254/13-07-2022Β
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Pain, Postoperative; Pain, Acute; Pain, Chronic; Pain, Nociceptive; Ketamine; Lidocaine; Analgesia; Analgesics; Cervical Spine Surgery
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chronic Pain; Nociceptive Pain; Agnosia | interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine-lidocaine (KL) group combination of ketamine and lidocaine in one syringe (Active Comparator)
  Interventions: Drug: ketamine-lidocaine
- : remifentanil group syringe of remifentanil (Active Comparator)
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: ketamine-lidocaine — In the KL group, patients will be administered in a total volume of 20 mL,1mL/10 kg of the solution containing ketamine, lidocaine at predefined concentrations.
  As maintenance, they will be receiving 1mL/10kg/h of the aforementioned solution
  Other Names: KL group
  Arms: ketamine-lidocaine (KL) group combination of ketamine and lidocaine in one syringe
Drug: Remifentanil — In the Remifentanil group, patients will be administered in a total volume of 20 mL, 2 mcg/kg of fentanyl. As maintenance, they will be receiving 1 mL/10kg/h of a remifentanil solution
  Other Names: Remifentanil group
  Arms: : remifentanil group syringe of remifentanil

SUMMARY:
The aim of this double blind randomized study will be to investigate the effect of an opioid-free anesthesia regimen with a mixture of lidocaine and ketamine in the same syringe versus remifentanyl analgesia in cervical spine surgery.

DETAILED DESCRIPTION:
Cervical spine surgery is associated with medium pain scores and perioperative disability. Ketamine and lidocaine have all proven but varied analgesic effects. High opioid consumption has been associated with multiple side effects.

This double blind clinical trial aims to investigate the possible reduction of opioid use during lumbar spine surgery by administering ketamine and lidocaine. Sixty patients will be randomly allocated into two groups. The control group will receive a continuous infusion of remifentanil, while the Ketamine-Lidocaine (KL) group will receive a continuous infusion of ketamine and lidocaine, during the surgery and shortly after.

Both infusions will be administered blindly. Fentanyl and morphine will be administered to each patient so as to maintain hemodynamic stability and pain relief. The study will eventually compare the need for bolus doses of fentanyl during the surgery and morphine shortly after in each group.

Multiple hemodynamic parameters, analgesic consumption, possible side effects, patient satisfaction and the Oswestry low back pain disability questionnaire will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adult patents
* American Society of Anesthesiologists (ASA) class I-III
* elective spine surgery

Exclusion Criteria:

* body mass index (BMI) >35 kg/m2
* contraindications to local anesthetic administration
* systematic use of analgesic agents preoperatively
* chronic pain syndromes preoperatively
* neurological or psychiatric disease on treatment
* pregnancy
* severe hepatic or renal disease
* history of cardiovascular diseases/ arrhythmias/ conduction abnormalities
* bradycardia(<55 beats/minute)
* drug or alcohol abuse
* language or communication barriers lack of informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
pain score on arrival to Post-Anesthesia Care Unit (PACU) | immediately postoperatively]
  pain score by the use of Numeric Rating Scale (NRS) on arrival to PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score at discharge from Post-Anesthesia Care Unit (PACU) | at discharge from Post Anesthesia Care Unit (PACU), approximately 1 hour postoperatively
  pain score by the use of Numeric Rating Scale (NRS) at discharge from PACU, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 3 hours postoperatively | 3 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 3 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 6 hours postoperatively | 6 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 6 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
pain score 24 hours postoperatively | 24 hours postoperatively
  pain score by the use of Numeric Rating Scale (NRS) 24 hours postoperatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"

SECONDARY OUTCOMES:
sedation on arrival to Post-Anesthesia Care Unit | immediately postoperatively
  sedation will be assessed with a 5-point sedation scale, where: 1, patient perfectly conscious; 2, patient feels a little drowsy; 3, patient seems to be sleeping but immediately reacts to verbal stimulation; 4, patient seems to be sleeping but slowly reacts to verbal stimulation and 5, patient seems to be sleeping and does not react to verbal stimulation but does react to a stimulus such as shaking or pain
sedation at discharge from Post-Anesthesia Care (PACU) Unit | at discharge from Post Anesthesia Care Unit (PACU), approximately 1 hour postoperatively
  sedation will be assessed with a 5-point sedation scale, where: 1, patient perfectly conscious; 2, patient feels a little drowsy; 3, patient seems to be sleeping but immediately reacts to verbal stimulation; 4, patient seems to be sleeping but slowly reacts to verbal stimulation and 5, patient seems to be sleeping and does not react to verbal stimulation but does react to a stimulus such as shaking or pain
time to first request for analgesia | during stay in Post-Anesthesia Care Unit (PACU), approximately 1 hour postoperatively
  the time for the first patient request for analgesia will be noted
morphine consumption in Post-Anesthesia Care Unit (PACU) | immediately postoperatively
  mg of morphine requested during patient PACU stay
tramadol consumption in the first 48 hours | 48 hours postoperatively
  patients will be followed for cumulative tramadol consumption for 48 hours postoperatively
fentanyl requirement during surgery | intraoperatively
  dose of required fentanyl intraoperatively to maintain systolic arterial blood pressure and heart rate within the 20% of baseline value
satisfaction from postoperative analgesia | 24 hours postoperatively
  satisfaction from postoperative analgesia on a six-point Likert scale with 1 marked as minimal satisfaction and 6 as maximal satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, Principal Investigator — Aretaieion University Hospital, Athens, Greece
Locations (1):
- Evangelismos General Hospital, Athens, Greece